CLINICAL TRIAL: NCT03458494
Title: The TCF7L2 Gene: Nutrigenomics and Dietary Prevention of Type 2 Diabetes
Brief Title: The TCF7L2 Gene: Dietary Prevention of T2DM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Tufts University (Other)
Collaborators: Allen Foundation Inc. (Other)
Responsible Party: Principal Investigator, Jose Ordovas, Senior Scientist, Lab Director JM-USDA-HNRCA, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: TCF7L2_2965
Record Dates: First submitted 2018-02-24; First posted 2018-03-08 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Type2 Diabetes; Glucose, High Blood
Keywords: type 2 diabetes; glucose; insulin; CRP; Metabolomics; gene-diet interaction; TCF7L2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Diet, Mediterranean; Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: randomized crossover dietary intervention
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet (Experimental): during one week participants will receive food products common in the diet of Mediterranean populations
  Interventions: Other: Mediterranean Diet
- Low-fat diet (Experimental): during one week participants will receive food products low in fat content
  Interventions: Other: Low-fat diet

INTERVENTIONS:
Other: Mediterranean Diet — Participants will receive meals traditionally consumed in Mediterranean countries
  Arms: Mediterranean Diet
Other: Low-fat diet — Participants will receive meals with a low content of total fat.
  Arms: Low-fat diet

SUMMARY:
Nutrients and chemicals in food are able to regulate expression of genetic elements. Gene-nutrient interaction in response specific diets can increase an individual's risk, shifting the individual from health toward the development of chronic disease. The Transcription Factor 7 Like 2 (TCF7L2) gene may either put individuals at risk for or protect from Type 2 diabetes mellitus in the presence of certain foods. The main purpose of this four-week study is to examine diet-induced gene-nutrient interaction, with a focus on glucose, insulin, inflammation (CRP) and the plasma metabolome in individuals who have either the CC or the TT form of the rs7903146 single nucleotide polymorphism (SNP) (C/T) within the TCF7L2 gene. The (2) one-week study diets, one Mediterranean diet (MedDiet) based and the other low-fat based will be separated by a (1) week return to a regular habitual diet.

DETAILED DESCRIPTION:
Type 2 diabetes (T2DM) is associated with increased morbidity and mortality, and its growing prevalence represents a major public health concern. T2D results from a combination of genetics and the exposure to external factors (i.e., diet, exercise, and stress). Multiple T2D-related genes have been identified, but they explain only ~10% of the estimated T2D heritability. Therefore, it has been proposed that interactions between genetic and environmental factors contribute to the missing heritability. The identification of these gene-environment interactions could provide a breakthrough in the prevention of T2D and its complications through the implementation of novel nutrigenomics approaches.

The rs7903146 single nucleotide polymorphism (SNP) (C/T) within the TCF7L2 gene is the most replicated T2D-associated SNP. However, the mechanism associating TCF7L2 with T2D remains unknown. Moreover, there is little knowledge of how diet modulates this association. A better understanding is crucial for improving existing, or designing new interventions for T2D prevention.

The current knowledge supports the notion that subjects homozygous for the deleterious allele (TT) have a higher risk of T2D than subjects homozygous for the common allele (CC). Furthermore, there is a gene-diet interaction between this SNP and Mediterranean diet (MedDiet) on fasting glucose and lipids. Thus, a higher MedDiet adherence neutralizes the effects of the deleterious TT genotype. Moreover, after ~5 years, TT subjects consuming a low-fat diet have higher incidence of stroke than CC subjects, whereas this association is annulled in TT subjects consuming a MedDiet. the objective of this study is to validate these findings under practical conditions similar to those encountered in clinical practice and to identify biological mechanisms involved in such interactions.

For this purpose, a four-week study will be conducted to examine diet-induced gene-nutrient interaction, with a focus on glucose, insulin, and inflammation (CRP) in individuals who have either the CC or the TT form of the rs7903146 single nucleotide polymorphism (SNP) (C/T) within the TCF7L2 gene. The (2) one-week study diets, one Mediterranean diet (MedDiet) based and the other low-fat based will be separated by a (1) week return to a regular habitual diet.

The specific aims include:

1. To investigate whether the TCF7L2-by-diet interaction in relation to T2D and cardiovascular disease (CVD) risk factors can be validated in the context of a more realistic scenario of personalized dietary advice based on genetic information (nutrigenomics).
2. To elucidate the molecular mechanisms responsible for these gene-by-diet interactions using deep phenotyping (i.e., metabolomics).

The hypothesis is that genetics can offer precise information about which healthy diet (low-fat or Mediterranean) can deliver real benefits on an individual basis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women.
* 18 years or older.
* Women who are not pregnant.
* A BMI ranging between 27 and 34

Exclusion Criteria:

* Unexplained elevation in serum transaminases (i.e. >1.5 times the upper limit of normal) or with evidence of active liver disease, including primary biliary cirrhosis or pre-existing gallbladder disease.
* Severe renal dysfunction (serum creatinine >2.0mg/dL).
* Excessive alcohol consumption (>2 drinks/day).
* Preexisting CVD.
* Stable exertional angina pectoris requiring sublingual nitroglycerin within the prior 3 months.
* Uncontrolled T2D (fasting glucose >126 mg/dl) or other significant endocrine disease.
* Uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg).
* History of pancreatitis within 1 yr. prior to screening.
* Subjects on lipid-lowering or diabetes medications.
* Smoking.
* Pregnancy.
* Body mass index (BMI) below 27 or greater than 34 kg/m2
* Participants will also be excluded for drug abuse, extreme dietary habits, multiple food allergies, extreme levels of physical or athletic activity, or by changes in body weight >20 lbs. during the last 6 months.
* Inability to follow any of the experimental diets or to perform the sampling required for this study.
* Thyroid diseases.
* Use of omega-3 supplements (unless it is discontinued one month prior to the beginning of the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Glucose | 1 week per intervention arm
  Plasma glucose levels (mg/dl) will be measured in the fasting state during each one of the intervention phases (the Mediterranean and low-fat diets) in participants with the TT and CC genotypes at the TCF7L2 rs7903146 SNP

SECONDARY OUTCOMES:
Insulin | 1 week per intervention arm
  Fasting plasma insulin levels (pmol/l) will be measured in the fasting state during each one of the intervention phases (the Mediterranean and low-fat diets) in participants with the TT and CC genotypes at the TCF7L2 rs7903146 SNP
Metabolomics | 1 week per intervention arm
  The response of plasma metabolites to the Mediterranean and low-fat diets diet) will be measured using ultra high-performance liquid chromatography/tandem accurate mass spectrometry (UHPLC/MS/MS) during each one of the intervention phases (the Mediterranean and low-fat diets) in participants with the TT and CC genotypes at the TCF7L2 rs7903146 SNP
Very low density lipoproteins (VLDL) | 1 week per intervention arm
  Fasting plasma concentrations of VLDL in mg/dl, assessed by proton nuclear magnetic resonance (NMR) spectroscopy will be measured during each one of the intervention phases (the Mediterranean and low-fat diets) in participants with the TT and CC genotypes at the TCF7L2 rs7903146 SNP
Low-density lipoproteins (LDL) | 1 week per intervention arm
  Fasting plasma concentrations of LDL in mg/dl, assessed by proton nuclear magnetic resonance (NMR) spectroscopy will be measured during each one of the intervention phases (the Mediterranean and low-fat diets) in participants with the TT and CC genotypes at the TCF7L2 rs7903146 SNP
High-density lipoproteins (HDL) | 1 week per intervention arm
  Fasting plasma concentrations of HDL in mg/dl, assessed by proton nuclear magnetic resonance (NMR) spectroscopy will be measured during each one of the intervention phases (the Mediterranean and low-fat diets) in participants with the TT and CC genotypes at the TCF7L2 rs7903146 SNP
CRP | 1 week per intervention arm
  Plasma C-reactive protein (mg/dl) will be measured in the fasting state during each one of the intervention phases (the Mediterranean and low-fat diets) in participants with the TT and CC genotypes at the TCF7L2 rs7903146 SNP

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Ordovas, PHD, Principal Investigator — Tufts University
Locations (1):
- JM-USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plans are in place to share individual participant data (IPD) with other researchers others than those involved in the study. However, the study investigators are open to collaborations that do not include sharing IPD

REFERENCES:
- [Background] Corella D, Carrasco P, Sorli JV, Estruch R, Rico-Sanz J, Martinez-Gonzalez MA, Salas-Salvado J, Covas MI, Coltell O, Aros F, Lapetra J, Serra-Majem L, Ruiz-Gutierrez V, Warnberg J, Fiol M, Pinto X, Ortega-Azorin C, Munoz MA, Martinez JA, Gomez-Gracia E, Gonzalez JI, Ros E, Ordovas JM. Mediterranean diet reduces the adverse effect of the TCF7L2-rs7903146 polymorphism on cardiovascular risk factors and stroke incidence: a randomized controlled trial in a high-cardiovascular-risk population. Diabetes Care. 2013 Nov;36(11):3803-11. doi: 10.2337/dc13-0955. Epub 2013 Aug 13. PMID 23942586
- [Derived] Lai CQ, Gervis JE, Parnell LD, Lichtenstein AH, Ordovas JM. Changes in triglyceride-rich lipoprotein particle profiles in response to one-week on a low fat or Mediterranean diet by TCF7L2 rs7903146 genotype: a randomized crossover dietary intervention trial. Genes Nutr. 2025 Mar 6;20(1):4. doi: 10.1186/s12263-025-00763-y. PMID 40050721